CLINICAL TRIAL: NCT00396825
Title: Phase II Trial of a Video That Presents Training in Stress Coping Skills for Caregivers of a Relative With Alzheimer's Disease or Other Dementia
Brief Title: Video-Based Coping Skills Training for Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Williams LifeSkills (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Virginia P. Williams, Ph.D., President, Williams LifeSkills
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2R44AG025593-04A;; 2R44AG025593 (NIH)
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Caregivers
Keywords: Care giving; Alzheimer's Disease; Stress management
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active treatment (Experimental): Subjects randomized to this arm will receive the Family Caregiver Kit composed of the Williams LifeSkills Family Caregiver Video and Workbook and will also receive telephone coaching
  Interventions: Behavioral: Video-based coping skills training with telephone coaching
- Control (No Intervention): Subjects randomized to this arm will receive no intervention and serve as wait list controls. They will undergo the same evaluations as the Intervention arm subjects at comparable times. In a crossover design, once subjects have finished serving as controls, they will be given the video, workbook, and telephone calls from a social worker and tested one more time.

INTERVENTIONS:
Behavioral: Video-based coping skills training with telephone coaching — Subjects will view the 10 modules of Williams LifeSkills Caregiver Video, do Workbook exercises for each module, and receive telephone coaching to enhance their ability to apply the skills taught in each module to caregiver situations.
  Other Names: Williams LifeSkills Family Caregiver Kit
  Arms: Active treatment

SUMMARY:
The purpose of this Phase II SBIR study is a) to complete the adaptation begun in Phase I of the ten skill modules of the Williams LifeSkills Video (WLV) for use by persons who are caregivers for a relative with Alzheimer's Disease (AD) or other dementia, b) to script and produce the complete Caregiver LifeSkills Video (CLV) and c) to conduct a randomized clinical trial of the completed CLV to document benefits in terms of reduced psychosocial distress, reduced biomarkers of stress and improved well being.

DETAILED DESCRIPTION:
An extensive body of research documents adverse effects of being a caregiver for a relative with AD on a broad range of psychosocial and biological indicators of stress, including increased hassles and depression (Russo & Vitaliano, Experimental Aging Research 1995; 21:273-294 ) and the metabolic syndrome (Vitaliano et al, Journal of Gerontology: Psychological Sciences 1996; 51:290-299). Interventions to reduce psychological distress in caregivers have not produced clinically meaningful results thus far (Shulz et al. Gerontologist 2002; 42:589-602) and no intervention trials have included assessment of biomarkers of stress. Logistic obstacles make it hard for caregivers to participate in treatments that require them to come to a treatment site outside the home; thus, interventions with caregivers are hard to deliver. The Williams LifeSkills Video (WLV) is based on the LifeSkills Workshop, which has been shown in randomized clinical trials to reduce hostility and blood pressure in post-MI patients (Gidron et al. Health Psychology 1999; 18:416-420) and to reduce a broad range of psychosocial risk factors as well as blood pressure and heart rate during both rest and stress conditions in post-CABG patients (Bishop et al., American Heart Journal 2005;150:602-609). The WLV was developed with support from an NIMH SBIR Phase II grant and presents 10 skill modules -- 1) increased awareness of thoughts and feelings arising in stressful situations; 2) evaluation of those thoughts and feelings to decide whether to try to change them or to take action to try to change the situation; 3) deflection skills to change one's thoughts and feelings; action skills to change stressful situations, including 4) assertion, 5) problem-solving, and 6) saying no; and relationship skills - 7) speaking clearly, 8) listening, 9) empathy, and 10) increasing the positives - using dramatizations of scenarios in which the skill is first not used and then used to produce a better outcome. A randomized clinical trial evaluating it in stressed community volunteers showed that it is superior to a wait list control condition in reducing psychosocial (anxiety, depression and perceived stress; (Kirby et al.Psychosomatic Medicine,2006;68:816-823.

In the research conducted in Phase I of this SBIR-supported study, we adapted the scenarios used for the 10 skills to represent more closely the real life situations faced by caregivers and we developed a telephone coaching manual. Now in Phase II of this study, we will produce the complete Caregiver LifeSkills Video (CLV) evaluate its effects on measures of psychosocial distress and biomarkers of stress in a randomized clinical trial with 120 caregivers of a relative with AD or other major dementias. If successful in reducing the psychosocial and biological markers of stress that are elevated in caregivers, this new WLS product, the CLV, could have a major impact in reducing the health damaging effects of stress among the millions of Americans who are caregivers for relatives with AD and other dementias.

ELIGIBILITY:
Inclusion Criteria:

* Must be a primary caregiver for a relative with Alzheimer's Disease or other dementia

Exclusion Criteria:

* Presence of a major medical or psychiatric illness that would prevent completion of low risk study procedures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiological Studies Depression scale | Pre- and post-training, 3 months and 6 months
Spielberger State-Trait Anger and Anxiety Scales | Pre-and post-training, 3 months and 6 months
Perceived Stress Scale | Pre- and post-training, 3 months and 6 months
Pittsburgh Sleep Quality Index | Pre-and post-training, 3 months and 6 months
Heart rate and blood pressure at rest and during recall of caregiver situation | Pre-and post-training, 3 months and 6 months
Salivary cortisol upon awakening, 30 minutes later, and prior to going to bed at night | Pre-and post-training, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Virginia P Williams, Ph.D., Principal Investigator — Williams LifeSkills
Locations (1):
- Williams LifeSkills, Inc., Durham, North Carolina, United States

REFERENCES:
- [Derived] Williams VP, Bishop-Fitzpatrick L, Lane JD, Gwyther LP, Ballard EL, Vendittelli AP, Hutchins TC, Williams RB. Video-based coping skills to reduce health risk and improve psychological and physical well-being in Alzheimer's disease family caregivers. Psychosom Med. 2010 Nov;72(9):897-904. doi: 10.1097/PSY.0b013e3181fc2d09. Epub 2010 Oct 26. PMID 20978227